CLINICAL TRIAL: NCT00020254
Title: A Randomized Phase II Study of Either Immunotherapy With a Regimen of Recombinant Pox Viruses That Express PSA/B7.1 Plus Adjuvant GM-CSF and IL2 or Hormone Therapy With Nilutamide in Patients With Hormone Refractory Prostate Cancer and No Radiographic Evidence of Disease
Brief Title: Vaccine Therapy Plus Sargramostim and Interleukin-2 Compared With Nilutamide Alone in Treating Patients With Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000068106; NCI-00-C-0137; MB-NAVY-99-04; NCI-T99-0097; NCT00005759 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2003-04

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — aldesleukin; PROSTVAC; sargramostim; nilutamide

INTERVENTIONS:
Biological: aldesleukin
Biological: recombinant fowlpox-prostate specific antigen vaccine
Biological: recombinant vaccinia prostate-specific antigen vaccine
Biological: recombinant vaccinia-B7.1 vaccine
Biological: sargramostim
Drug: nilutamide

SUMMARY:
RATIONALE: Vaccines made from prostate cancer cells may make the body build an immune response to kill tumor cells. Colony-stimulating factors such as sargramostim may increase the number of immune cells found in bone marrow or peripheral blood. Interleukin-2 may stimulate a person's white blood cells to kill prostate cancer cells. Androgens can stimulate the growth of prostate cancer cells. Hormone therapy using nilutamide may fight prostate cancer by reducing the production of androgens. It is not yet known which treatment regimen is more effective for treating prostate cancer.

PURPOSE: Randomized phase II trial to compare the effectiveness of vaccine therapy plus sargramostim and interleukin-2 with that of nilutamide alone in treating patients who have prostate cancer that has not responded to hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the difference in time to radiographic evidence of disease progression at 6 months in patients with hormone-refractory prostate cancer when treated with vaccine containing recombinant vaccinia-prostate-specific antigen (PSA) admixed with rV-B7.1 plus recombinant fowlpox-PSA vaccine, sargramostim (GM-CSF), and interleukin-2 vs nilutamide alone.
* Evaluate the vaccination therapy in relation to the change in T-cell precursor frequency and to the rise of serum PSA in this patient population.

OUTLINE: This is a randomized study. Patients are stratified according to HLA-A2 typing (positive vs negative). Patients are randomized to one of two treatment arms.

* Arm I: Patients receive vaccine containing recombinant vaccinia-prostate-specific antigen (PSA) and rV-B7.1 subcutaneously (SC) on day 2 only. Beginning on day 30, patients receive recombinant fowlpox-PSA vaccine SC every 4 weeks for 12 vaccinations and then every 12 weeks thereafter. Patients also receive sargramostim (GM-CSF) SC daily on days 1-4 and interleukin-2 SC daily on days 8-12 with each vaccination.

Patients without disease progression after 12 courses receive the vaccine regimen every 12 weeks.

* Arm II: Patients receive oral nilutamide daily. Treatment continues in both arms for at least 6 months in the absence of disease progression or unacceptable toxicity.

After 6 months of therapy, patients with a rising PSA and no radiographic evidence of disease progression may receive therapy in the other arm in addition to the therapy to which they were randomized.

Patients are followed monthly for 6 months and then every 2 months thereafter.

PROJECTED ACCRUAL: A total of 56-78 patients (28-39 per treatment arm) will be accrued for this study within 1.5-2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed hormone-refractory adenocarcinoma of the prostate

  * Rising PSA after orchiectomy and/or while receiving at least 1 regimen of luteinizing hormone-releasing hormone (LHRH)
  * PSA must have risen at least 0.5 ng/mL from baseline on 2 successive measurements during and/or after hormonal therapy
  * PSA greater than 1.0 ng/mL
  * If on antiandrogen therapy, must undergo antiandrogen withdrawal for at least 6 weeks and still have evidence of rising PSA
  * After prior bicalutamide, must undergo withdrawal for at least 6 weeks and still have evidence of rising PSA
* Testosterone no greater than 50 ng/mL if no prior orchiectomy
* No metastatic disease by bone scan and CT scan or MRI of the abdomen and pelvis and by CT scan or x-ray of the chest
* No active or prior CNS metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Zubrod 0-2 OR
* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute lymphocyte count at least 600/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 8.0 g/dL

Hepatic:

* Bilirubin no greater than 1.6 mg/dL
* AST and ALT no greater than 4 times normal

Renal:

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance greater than 60 mL/min
* Urinalysis normal OR
* Proteinuria no greater than 1 g/24-hour urine collection
* No hematuria or abnormal sediment unless underlying cause is nonrenal

Immunologic:

* HIV negative
* No altered immune function
* No autoimmune disease, including the following:

  * Autoimmune neutropenia, thrombocytopenia, or hemolytic anemia
  * Systemic lupus erythematosus, Sjogren's syndrome, or scleroderma
  * Myasthenia gravis
  * Goodpasture syndrome
  * Addison's disease, Hashimoto's thyroiditis, or active Graves' disease
* No known allergy or untoward reaction to prior vaccination with vaccinia virus
* No known allergy to eggs
* No active or prior eczema or other eczematoid skin disorders
* No other acute, chronic, or exfoliative skin conditions (e.g., atopic dermatitis, impetigo, varicella zoster, burns, severe acne, or other open rashes or wounds)

Other:

* No other serious concurrent illness
* No active infections within the past 3 days
* No history of seizures, encephalitis, or multiple sclerosis
* No close or household contact for at least 2 weeks after each vaccinia virus inoculation with the following high-risk individuals:

  * Children under 5 years of age
  * Pregnant or nursing women
  * Individuals with active or prior eczema or other eczematoid skin disorders, atopic dermatitis, impetigo, varicella zoster, burns, severe acne, or other open rashes or wounds
  * Immunosuppressed or immunodeficient (by disease or therapy) individuals, including those with HIV infection
* No other malignancy within the past 3 years except squamous cell or basal cell skin cancer or other curatively treated malignancy

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Must have prior vaccinia for smallpox immunization
* No other concurrent biologic therapy

Chemotherapy:

* No prior chemotherapy for prostate cancer
* No concurrent chemotherapy

Endocrine therapy:

* See Disease Characteristics
* At least 4 weeks since prior hormonal therapy (6 weeks for bicalutamide) and recovered
* If disease progression on LHRH antagonist, must continue to receive that LHRH agent or undergo surgical castration
* No concurrent steroids unless topical or inhaled
* No other concurrent hormonal therapy

Radiotherapy:

* At least 4 weeks since prior radiotherapy and recovered
* No prior radiotherapy to more than 50% of nodal groups
* No concurrent radiotherapy

Surgery:

* See Disease Characteristics
* See Endocrine therapy
* At least 4 weeks since prior surgery and recovered
* No prior splenectomy

Other:

* No concurrent homeopathic therapy with PC-SPES or genistein

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-06; Primary Completion 2004-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip M. Arlen, MD, Study Chair — National Cancer Institute (NCI)
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland, United States

REFERENCES:
- [Background] Tsang KY, Zhu M, Even J, Gulley J, Arlen P, Schlom J. The infection of human dendritic cells with recombinant avipox vectors expressing a costimulatory molecule transgene (CD80) to enhance the activation of antigen-specific cytolytic T cells. Cancer Res. 2001 Oct 15;61(20):7568-76. PMID 11606396
- [Result] Madan RA, Gulley JL, Schlom J, Steinberg SM, Liewehr DJ, Dahut WL, Arlen PM. Analysis of overall survival in patients with nonmetastatic castration-resistant prostate cancer treated with vaccine, nilutamide, and combination therapy. Clin Cancer Res. 2008 Jul 15;14(14):4526-31. doi: 10.1158/1078-0432.CCR-07-5048. PMID 18628467
- [Result] Arlen PM, Gulley JL, Todd N, Lieberman R, Steinberg SM, Morin S, Bastian A, Marte J, Tsang KY, Beetham P, Grosenbach DW, Schlom J, Dahut W. Antiandrogen, vaccine and combination therapy in patients with nonmetastatic hormone refractory prostate cancer. J Urol. 2005 Aug;174(2):539-46. doi: 10.1097/01.ju.0000165159.33772.5b. PMID 16006888
- [Result] Arlen PM, Gulley JL, Novik L, et al.: A randomized phase II trial of either vaccine therapy (recombinant pox viruses expressing PSA and the B7.1 costimulatory molecule) versus hormone therapy (nilutamide) in patients with hormone refractory prostate cancer and no radiographic evidence of disease. [Abstract] J Urol 169 (4 Suppl): A-941, 243, 2003.
- [Result] Arlen PM, Gulley J, Novik L, et al.: A randomized phase II trial of either vaccine therapy (recombinant pox viruses expressing PSA and the B7.1 costimulatory molecule) versus hormone therapy (nilutamide) in patients (pts) with hormone refractory prostate cancer and no radiographic evidence of disease. [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-728, 2002.